CLINICAL TRIAL: NCT03349541
Title: A Multicenter Randomized Trial of Curricular Modules in the Care of Children With Medical Complexity for Paediatric Residents
Brief Title: Paediatric Resident Complex Care Curriculum RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other); Montreal Children's Hospital of the MUHC (Other)
Responsible Party: Principal Investigator, Julia Orkin, Staff Physician, Medical Director of the Complex Care Program, Project Investigator, SickKids Research Institute, Assistant Professor, Department of Pediatrics, University of Toronto, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1000056104
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Complex Care; Medical Education; Pediatric Residents; Children With Medical Complexity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex Care Curriculum Intervention (Experimental): Paediatric residents who are randomized to the intervention group will participate in the complex care curriculum during an academic half-day prior to the Objective Structured Clinical Examination (OSCE).
  Interventions: Other: Complex Care Curriculum
- No intervention (No Intervention): Paediatric residents who are randomized to the control group will attend the regular academic half-day unrelated to complex care prior to the Objective Structured Clinical Examination (OSCE).

INTERVENTIONS:
Other: Complex Care Curriculum — A well-established approach to curriculum development was utilized to develop competency-based objectives aligned with the Canadian "CanMEDS" Physician Competency Framework, identify appropriate educational strategies and design relevant evaluations.
  Arms: Complex Care Curriculum Intervention

SUMMARY:
Medical and technological advances have resulted in a growing cohort of children with medical complexity (CMC), many of whom would not have survived previously and are living and thriving within the community. These families have unique needs that have previously not been taught in the typical training programs for paediatricians. The goal of this project is to develop an evaluation of a national complex care curriculum and to identify whether dedicated educational modules have an impact on improving clinical performance and resident self-efficacy.

DETAILED DESCRIPTION:
Rationale:

A structured program evaluation considering a hierarchy of outcomes is essential to determine whether improved training in complex care is associated with increased skills in this area, and whether these skills transfer to a clinical setting where they will influence quality of care for CMC.

A paediatric resident's sense of self-efficacy, or perceived capability, in caring for CMC is therefore important to foster for the graduating paediatrician to assume a leadership role in coordinating care, co-developing goals of care with families, advocating in the face of health challenges, and ultimately striving for high-quality clinical care for CMC.

We anticipate that participation in a complex care curriculum will result in sustained high performance on simulated clinical scenarios in complex care and increased resident self-efficacy in caring for CMC, compared to paediatric residents that have not participated in the curriculum. This study will examine if a standardized complex care curriculum for paediatric residents has a positive effect on the acquisition of key competencies in the care of CMC using a rigorous experimental research design. To our knowledge, this is the first national, standardized, population-specific curriculum for Canadian paediatric residents to be developed and evaluated with this systematic approach.

Study Objectives:

The overarching aim of this project is to develop a robust evaluation of the national complex care curriculum, and identify whether dedicated educational modules have an impact on improving clinical performance and resident self-efficacy.

Primary Research Question:

What is the comparative effectiveness of participation in a standardized curriculum on acquisition of clinical skills in complex care for paediatric residents, relative to paediatric residents receiving a standard educational session not related to complex care, evaluated by OSCE scores in a complex care scenario?

Secondary Objectives:

To explore changes in paediatric residents' sense of self-efficacy and comfort in caring for CMC following participation in the curriculum using semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Residents in their 1st to 4th postgraduate year of training in paediatrics (general paediatric stream and paediatric neurology stream who have regular attendance at the academic half-days), enrolled at the University of Toronto or the University of Ottawa.

Exclusion Criteria:

* Residents who are enrolled in a subspecialty residency training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Acquisition of clinical skills in Complex Care | Within 1-3 months from complex care educational training (day of the scheduled OSCE examination)
  This outcome will be measured by the score obtained on a standardized checklist for a complex care scenario in the Spring 2017 national paediatric in-training objective structured clinical examination (OSCE). The OSCE global score is out of 50, with a higher score representing a better performance. OSCE sub-scores related to specific components of the curriculum (tracheostomy care, common issues in complex medical care, and diagnosis and management) will be compared between groups.

SECONDARY OUTCOMES:
Resident self-efficacy in the care of Children with Medical Complexity | Within 4 months from the complex care educational training
  This outcome will be explored through in-depth qualitative interviews.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No